CLINICAL TRIAL: NCT02378818
Title: SCHIZOBAT/DEPBAT : Characterization of the Motivational Deficit in Schizophrenia and Depression
Brief Title: Characterization of the Motivational Deficit in Schizophrenia and Depression
Acronym: SCHIZOBAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Institut du Cerveau et de la Moelle (ICM Institute) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D14-P012
Record Dates: First submitted 2014-08-13; First posted 2015-03-04 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia; Depression
Keywords: Schizophrenia; Negative symptoms; Lack of motivation; Cognitive characterization; Computational psychiatry; Depression
MeSH Terms: conditions — Schizophrenia; Depression | interventions — Advisory Committees

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Schizophrenia patients (Other): 35 patients, Age between 18 and 65 years, with a diagnosis of schizophrenia and unchanged psychotropic treatment for at least three months before inclusion.
  Interventions: Behavioral: Force task, preference task, discount task, learning task.
- Healthy volunteers (schizophrenia) (Other): 35 healthy volunteers
  Interventions: Behavioral: Force task, preference task, discount task, learning task.
- Depressive patients (Other)
  Interventions: Behavioral: Force task, preference task, discount task, learning task.
- Healthy volunteers (depression) (Other)
  Interventions: Behavioral: Force task, preference task, discount task, learning task.

INTERVENTIONS:
Behavioral: Force task, preference task, discount task, learning task. — Force task, preference task, discount task, learning task.

SUMMARY:
This research focuses on disorders of motivation, responsible for a disability that patients experience daily. It is a disorder that affects behavior, especially social. Mechanisms, which result in these disorders, are poorly understood. This ignorance is responsible for the lack of effective therapy. The investigators realize this work in order to better understand the motivational deficits. The objective of the study is to characterize the cognitive mechanisms of motivational deficits in schizophrenia and depression. To answer the question posed in the research, it is planned to include 35 people with schizophrenia, 35 people with depression and 70 heathy volunteers in the Hospital of Sainte-Anne .

DETAILED DESCRIPTION:
The investigator goal is to develop a neuropsychological battery to characterize the different aspects of motivation: energizing action, ability to use the clues to assign value, ability to anticipate a reward delayed in time, and finally learning by trial / error based rewards. In addition, the investigators systematically compare the effect of rewards and punishments (losses) in these spots. Such a systematic approach should better understand the nature of disrupted in schizophrenia process. It should also highlight the differential effects of treatment, including the effects of conventional antipsychotics versus atypical antipsychotics, but also the benefits of cognitive remediation.

In the depression:

The motivational deficit is at the heart of the depressive symptomatology. Our objective is to characterize the motivational processes altered in the depression thanks to the same neuropsychological battery. Furthermore, this clinical dimension could influence the answer to the antidepressant treatment. A better characterization of the motivational deficit would allow to adapt at best the pharmacological treatments used in the depression, in particular by targeting the dopaminergic way, involved in the control of the motivation.

The investigators will recruit 35 patients and 35 control subjects in both populations. The investigators will make them pass a battery of motivational tests described above on three half-days:

- Force task: This task tests the energization process, that is to say the ability to activate an action in proportion to what is involved.

It consists of two sessions of 60 trials, which are offset through six levels of monetary issue (1, 20, 50 cents, 1, 5, 20 euros), and lasts about 30 minutes. On each trial, patients must tighten the grip dynamometer in order to earn a reward proportional to both the level of monetary issue and the peak forces occurs, or avoid a financial loss of a magnitude equal. The award of this task will be made in subliminal conditions and in supraliminal, and in condition of mental effort with the use of a stroop test instead of the dynamometer.

- Preference task: This task tests the integrity of the "brain recovery system." It includes three subtests quotes 24 awards, 24 penalties and 24 efforts, and three subtests of binary choices with 48 trials each, and lasts about 30 minutes. Patients should note how various awards seem pleasant, how various punishments seem unpleasant, or how various efforts seem harsh. Registration vegetative markers (heart rate) compares the implied valuations for explicit assessments (notes), and thus to estimate the accuracy of introspection.

- Discount and effort task: These tasks are used to estimate the parameters of time counting efforts and punishments. In the task of counting time effort, patients must choose between making a small reward associated with a low time or earn a greater reward associated with a significant delay. In the task of temporal punishments count, patients must choose between experience low punishment in a short time, or suffer a greater punishment in a larger delay. These tasks can capture a form of apathy characterized by an exaggeration of fatigue or pain early.

- Learning task: It can test the overall learning abilities and specific sensitivities learning by positive and negative reinforcement. It consists of two sessions, each with 60 binary choices (24 associated with rewards, punishments associated with 24, 12 associated with neutral events), for a period of about 20 minutes. The second session will be provided in counterfactual condition.

ELIGIBILITY:
Inclusion Criteria (schizophrenia group) :

* Patients :

  * Age between 18 and 65 years
  * Affiliation to a healthy insurance
  * Subjects who were informed and willing to sign the form of free and informed consent and information of the curator if necessary (or consent of the tutor)
  * French native tongue
  * Diagnosis of schizophrenia according to ICD-10, made by a psychiatrist. The subjects are stabilized (less than three items include a score> = 4 or to the positive level (P) of the PANSS)
  * Unchanged psychotropic treatment for at least three months before inclusion, a minimal dose adjustment in the last month is tolerable.
* Healthy volunteers:

  * Age between 18 and 65 years
  * Affiliation to a healthy insurance
  * Subjects who were informed and willing to sign the form of free and informed consent and information curator appropriate
  * French native tongue

Exclusion Criteria (schizophrenia group) :

* Patients:

  * Unable major, persons deprived of liberty, pregnant women
  * Enforced hospitalisation
  * Recent abuse (1 week) or chronic use of addictive substances, except tobacco
  * Treatment electro-convulsivo-therapy in the last 6 months
  * Degenerative Pathology, neurological disorder
  * Co-occurrence of a major depressive episode in a schizophrenic patient evaluated by a score> 10 CDS
  * Difficulty in understanding and expression in French language
  * Deficit of visual acuity or uncorrected hearing
* Healthy volunteers:

  * Unable major, persons deprived of liberty, pregnant women
  * Current psychiatric disease
  * Psychotropic treatment
  * Recent abuse (1 week) or chronic use of addictive substances, except tobacco
  * Difficulty in understanding and expression in French language
  * Deficit of visual acuity or uncorrected hearing
  * Mental retardation

Inclusion Criteria (depression group) :

* Patients :

  * Age between 18 and 75 years
  * Affiliation to a healthy insurance
  * Subjects informing and accepting to sign the free and lit consent form and information of the curator if necessary or consent of the tutor
  * French Mother tongue
  * Diagnosis of major depressive episode following the CIM-10, put by a psychiatrist.
* Healthy volunteers:

  * age between 18 and 75 years
  * Affiliation to a healthy insurance
  * Subjects informing and accepting to sign the free and lit consent form
  * French mother tongue

Exclusion Criteria (depression group) :

* Patients

  * persons deprived of liberty , pregnant women
  * Admission under constraint
  * Recent Abuse ( 1 week) or consumption chronicles of addicting substances, except the tobacco
  * Treatment by electroconvulsivo-therapy
  * Degenerative Pathology or obvious neurological disorder
  * Diagnosis of schizophrenia or disorder of personality severe
  * Difficulties of understanding and expression in French language
  * Uncorrected visual or hearing Deficit of acuteness
* Healthy volunteers:

  * Incapable, persons deprived of liberty, pregnant women
  * Recent Abuse (1 week) or consumption chronicles of addicting substances, except tobacco
  * Personal psychiatric Histories
  * Current psychiatric Disorder
  * Current psychotropic Treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-11-21 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
level of force produced based in incentive reward | the first inclusion day
level of force produced based in incentive reward | up to third day

SECONDARY OUTCOMES:
consistent level of choice questionnaire | the first inclusion day
The proportion of choosing the expensive option (great effort/big time/immediate effort) | the first inclusion day
The proportion of corrects choice | the first inclusion day

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël GAILLARD, MD, PhD, Principal Investigator — Centre Hospitalier St Anne
Locations (1):
- Centre Hospitalier Sainte Anne, Paris, France